CLINICAL TRIAL: NCT02640742
Title: Asthma Control, Quality of Life and Emotional Feelings in a Real Life Setting-A Cross-sectional Study of Adult Asthma Patients in Japan
Brief Title: Asthma Control, Quality of Life and Emotional Feelings in a Real Life Setting
Acronym: ACQUIRE-2
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00101
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate the asthma control status, asthma symptoms (severity, frequency, and limitations on activities, etc.), QOL, and use of drugs for asthma attack in adult asthma patients.

DETAILED DESCRIPTION:
Rationale for this Non-Interventional Study According to the Japanese Asthma Prevention and Management Guideline 2015 (Japan guideline (JGL) 2015), the goal in the management and treatment of asthma is "to be able to lead a life like a healthy individual." In order to achieve this therapeutic goal, the achievement of "well-controlled" state based on the asthma control status is considered to be a clinical goal. However, there are few studies in which the asthma control status is accurately surveyed in a real life setting in adult asthma patients receiving continued treatment from physician in Japan and the actual situation is unknown. By understanding the status of asthma control in asthma patients in a real life setting, the clinical issues could be clarified. Therefore, such information would contribute to appropriate treatment of asthma.

Thus, we planned this study to evaluate the asthma control status, asthma symptoms (severity, frequency, and limitations on activities, etc.), Quality of line (QOL), and use of drugs for asthma attack in the study population in a real life setting by recruiting patients through medical institutions providing continued care for asthma patients.

Objectives of this Non-Interventional Study

1. Primary objective

   To assess the proportion of adult asthma patients receiving continued treatment from physician in Japan in each asthma control status defined by JGL 2015 ("poorly-controlled," "insufficiently-controlled," and "well-controlled").
2. Secondary objectives

To evaluate asthma symptoms (intensity, frequency, and limitations on activities, etc.), QOL, use of drugs for asthma attack, and emotional feelings in the study population; and to investigate the effects of demographic characteristics and pathologic properties of each patient on the status of asthma control, asthma symptoms, QOL, use of drugs for asthma attack, and emotional feelings.

ELIGIBILITY:
Inclusion Criteria:

* Provided written consent before starting any procedure specified in the study protocol
* Aged 20 years or older at the time of providing the consent
* Receiving treatment for asthma as an outpatient at the time of providing the consent
* Physician definitive diagnosis of asthma at least 1 year before providing the consent
* Started to receive treatment with at least 1 of the following asthma drugs at least 1 year before providing the consent

Exclusion Criteria:

* Enrolled in this study in the past
* Assessed by the Investigator to require additional treatment due to worsening of asthma symptoms at the time of providing the consentEnrolled in this study in the past
* Scheduled to be hospitalized within 2 weeks after providing the consent due to asthma or any other disease
* Participating in another interventional study such as a clinical study at the time of providing the consent
* Considered by the Investigator as not appropriate for enrollment in this study due to inability to adhere to the procedures, limitations, and requirements of this study including answering and returning the questionnaires, etc.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult asthma patients receiving continued treatment by physician in Japan
Sampling Method: Non-Probability Sample
Enrollment: 1232 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
The primary variable is status of asthma control in each patient | Day1 to Day7
  Status of asthma control will be evaluated based on the patient diary and information in the clinical report form (CRF). Of the 6 items of Japanese guideline(JGL) 2015, the following 4 items will be used as indicators for evaluation of asthma control status: asthma symptoms (daytime and nighttime), use of a drug for asthma attack, limitation on activities including exercise, exacerbation (unscheduled visit, emergency room visit, and hospitalization).
  Status of asthma control in each patient ("well controlled," "insufficiently controlled," and "poorly-controlled" ) will be evaluated according to the evaluation criteria in JGL 2015.

SECONDARY OUTCOMES:
Asthma symptoms | Baseline
  To be evaluated based on Patient diary.
Use of drugs for the treatment of asthma | Baseline
  To be evaluated from case report form.
Asthma control during the past 1 week | Baseline
  To be evaluated by Asthma Control Questionare-5 (Japanese Version).
Asthma control status during the past 1 month | Baseline
  To be evaluated based on Patients' Questionnaire, case report form.
QOL | Baseline
  To be evaluated by Mini Asthma Quality of Life Questionnaire (Japanese Version)
Use of drugs for asthma attack and emotional feelings | Baseline
  To be evaluated based on Patients' Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Adachi, MD, PhD, Professor, Principal Investigator — International University of Health and Welfare; Gen Tamura, MD, PhD, President, Principal Investigator — Airway Institute in Sendai Co., Ltd; Masanori Nishikawa, DM, PhD, Principal Investigator — Department of Respiratory Medicine, Fujisawa City Hospital; Soichiro Hozawa, MD, Principal Investigator — Hiroshima Allergy and Respiratory Clinic
Locations (57):
- Japan (57):
  - Hiramatsu Clinic, Specializing in Internal Medicine, Respiratory Internal Medicine, Asthma, Sleep and Total Care of Rehabilitation in Respiratory in Komaki, Komaki, Aichi-ken
  - Toyota Memorial Hospital, Toyota, Aichi-ken
  - Ken Respiratory & Allergy Clinic, Hachinohe, Aomori
  - Fukuokaken Saiseikai Futsukaichi Hospital, Chikushino-shi, Fukuoka
  - Japan Community Health Care Organization Kurume General Hospital, Kurume, Fukuoka
  - Kumashiro Hospital, Kurume, Fukuoka
  - Ikedo Cardiovascular Medicine Clinic, Kurume, Fukuoka
  - Omuta Tenryo Hospital, Omuta, Fukuoka
  - Omuta Hospital, Omuta, Fukuoka
  - Takagi Hospital, Ōkawa, Fukuoka
  - Nagata Hospital, Yanagawa, Fukuoka
  - Fujita General Hospital, Date-gun, Fukushima
  - Tohno Chuo Clinic, Mizunami, Gifu
  - Tsuchiya Clinic, Takasaki, Gunma
  - Idaimae Minami Yojo Naika Clinic, Sapporo, Hokkaido
  - Nakatani Hospital, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital, Kobe, Hyōgo
  - Sudo Clinic, Morioka, Iwate
  - Sakaide City Hospital, Sakaidechō, Kagawa-ken
  - Takamatsu Hospital, Takamatsu, Kagawa-ken
  - Kamei Internal Medicine & Respiratory Clinic, Takamatsu, Kagawa-ken
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Furuie Clinic, Yokohama, Kanagawa
  - Saiseikai Yokohama Southern Hospital, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - National Hospital Organization Fukuoka-Higashi Medical Center, Fukuoka, Koga
  - Sendai Medical Center, Sendai, Miyagi
  - National Hospital Organization Minami-Okayama Medical Center, Tsukubo-gun, Okayama-ken
  - Kawaguchi Respiratory Medicine Clinic, Higashiosaka, Osaka
  - Ikeda City Hospital, Ikeda, Osaka
  - Matsushita Memorial Hospital, Moriguchi, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Takatsuki General Hospital, Takatsuki, Osaka
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - Iwata City Hospital, Iwata, Shizuoka
  - Nihonbashi Medical & Allergy Clinic, Cyuo-ku, Tokyo
  - Futaba-cho Clinic, Itabashi-ku, Tokyo
  - National Hospital Organization Tokyo National Hospital, Kiyose, Tokyo
  - Yamazaki Chest Clinic, Koganei, Tokyo
  - Jinyu Clinic Hospital, Nakano-ku, Tokyo
  - Senzoku Kokyuuki & Allergy Clinic, Ōta-ku, Tokyo
  - National Center for Global Health and Medicine, Shinjyuku-ku, Tokyo
  - The Fraternity Memorial Hospital, Sumida-ku, Tokyo
  - Yuizen Clinic, Tachikawa, Tokyo
  - Hamanomachi Hospital, Fukuoka
  - Fukuoka Sanno Hospital, Fukuoka
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka
  - Ohara General Hospital, Fukushima
  - Sakurai Clinic, Hiroshima
  - Hiroshima Allergic & Respiratory Clinic, Hiroshima
  - Tsuya Internal Medicine & Respiratory Department Clinic, Hiroshima
  - Yodogawa Christian Hospital, Osaka
  - Saga-ken Medical Centre Koseikan, Saga
  - Saitama Red Cross Hospital, Saitama
  - Shizuoka General Hospital, Shizuoka

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4064&filename=ACQUIRE-2_CSR_Synopsis_v1-0‗20171019.pdf